CLINICAL TRIAL: NCT00352339
Title: Switch Risperidone to Aripiprazole in Early Stage of Pharmacotherapy of Schizophrenia
Brief Title: The New Strategy for Pharmacological Treatment in People With Schizophrenia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inje University (Other)
Responsible Party: Busan Paik Hospital, Inje University, Clinical Trial Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Aripiprazole study 2006
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2009-08-06 (Estimated); Status verified 2009-08

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Switching; Early stage; Risperidone; Aripirazole
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Aripiprazole (Experimental): switching group (from risperidone to aripiprazole)
  Interventions: Drug: Rispridoen and Aripiprazole
- Risperidone (Active Comparator): Start with risperidone and keep it through the end of study
  Interventions: Drug: Risperidne
- Abilify (Active Comparator): Start with aripiprazole and keep it through the end of study
  Interventions: Drug: Abilify

INTERVENTIONS:
Drug: Rispridoen and Aripiprazole — Start with risperidone and switch it to aripiprazole. Flexible dose
  Arms: Aripiprazole
Drug: Risperidne — Start with risperidne and keep it through the end of study. Risperidne:flexible dose
  Arms: Risperidone
Drug: Abilify — Start with abilify and keep it through the end of study
  Other Names: abilify is a generic name of aripiprazole
  Arms: Abilify

SUMMARY:
Switching from Risperidone to Aripiprazole in early stage of pharmacotherapy will demonstrate the same efficacy as compared to risperidone continuation treatment in the treatment of schizophrenia.

DETAILED DESCRIPTION:
It has been thought that D2 Blocking agent is necessary in acute as well as maintenance phase of pharmacological treatment of patients with schizophrenia. However, this classical strategy produces long term adverse events of drug such as TD, osteoporosis and some metabolic syndrome. To overcome these adverse events, new strategy for pharmacological treatment is needed.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia, DSM-IV
* Acute phase

Exclusion Criteria:

* Refractory Schizophrenia
* Substance Abuse
* High risk for suicide

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
SANS(Scale for the Assessment of Negative Symptoms) | 12 weeks

SECONDARY OUTCOMES:
SARS(Simpson-Angus Rating Scale) | 12 weeks
Drug Attitude Inventory | 12 weeks
Side effect checklist | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Cheol Shim, MD,PhD, Principal Investigator — Clinical Trial Center, Paik hospital
Locations (2):
- South Korea (2):
  - Dongrae Hospital, Busan
  - Dongseo Hospital, Masan